CLINICAL TRIAL: NCT01451827
Title: A Phase 2, Multicenter, Randomized, Placebo-controlled, Double-blind, Placebo-masked, Parallel-group Pilot Trial to Compare the Efficacy, Tolerability, and Safety of Tolvaptan Modified-release and Immediate-release Formulations in Subjects With Autosomal Dominant Polycystic Kidney Disease
Brief Title: 8-Week Study of Tolvaptan Dose Forms in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Acronym: NOCTURNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 156-09-290
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Kidney Disease; Polycystic Kidney Disease; Autosomal Dominant Polycystic Kidney Disease; PKD; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases; Polycystic Kidney Diseases | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tolvaptan MR 50 mg (Experimental): Tolvaptan MR 50 mg capsule and 2 placebo IR tablets ( 8 AM) and 1 placebo IR tablet (4 PM) daily.
  Interventions: Drug: Tolvaptan MR; Drug: Placebo
- Tolvaptan MR 80 mg (Experimental): Tolvaptan MR 80 mg capsule and 2 placebo IR tablets (8 AM) and 1 placebo IR tablet (4 PM) daily.
  Interventions: Drug: Tolvaptan MR; Drug: Placebo
- Tolvaptan IR 60/30 mg (Experimental): Two tolvaptan IR 30-mg tablets and 1 placebo MR capsule (8 AM) and 1 tolvaptan IR 30-mg tablet (4 PM) daily.
  Interventions: Drug: Tolvaptan IR; Drug: Placebo
- Placebo (Placebo Comparator): Placebo MR capsule and 2 placebo IR tablets (8 AM) and 1 placebo IR tablet (4 PM) daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan MR — 50/80 mg capsules
  Other Names: OPC-41061
  Arms: Tolvaptan MR 50 mg; Tolvaptan MR 80 mg
Drug: Tolvaptan IR — 60/30 mg capsules
  Other Names: OPC-41061
  Arms: Tolvaptan IR 60/30 mg
Drug: Placebo — tablet

SUMMARY:
The purpose of this study is to compare the short-term effects of two tolvaptan formulations in patients with ADPKD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50
2. Subjects with:

   * BMI between 19 and 35 kg/m2
   * diagnosis of ADPKD by modified Ravine criteria:

     * family history: 3cysts/kidney if by sonography or 5 by CT or MRI
     * Without family history: 10 cysts per kidney
   * an eGFR > 45 mL/min/1.73 m2 by the CKD-EPI equation
3. Subjects not planning to become pregnant willing to comply with birth control requirements.
4. Subjects must be in good health as determined by screening tests.
5. Subjects providing informed consent and able to comply with all trial requirements.

Exclusion Criteria:

1. Subjects using diuretics within 14 days prior to randomization, or the requirement for intermittent or constant diuretic use for any reason
2. Subjects who had an eGFR < 45 mL/min/1.73 m2 calculated based on the most recent historical creatinine during the last 12 months
3. Subjects with:

   * incontinence, overactive bladder, or urinary retention (eg, BPH), meaning subjects with symptoms of frequent nocturia, as determined by medical history or urinary urgency should be carefully evaluated to exclude non-ADPKD GU issues prior to entry.
   * liver disease, liver function abnormalities, or serology other than that expected for ADPKD with cystic liver disease at baseline
   * a history of renal surgery or cyst drainage within 6 months of randomization
   * blood pressure 150/95 mmHg or < 90/40 mmHg.
   * heart rate outside the range of 40 to 90 bpm.
   * advanced diabetes with a history of poor control, evidence of significant renal disease renal cancer, single kidney, or recent renal surgery
   * other significant medical history that may interfere with the study objectives
   * significant abnormalities in serum sodium concentration (< 135 or > 145 mEq/L)
   * a history of drug and/or alcohol abuse within 2 years prior to screening
   * clinically significant allergic reactions to tolvaptan or chemically related structures such as benzazepines (eg, benzazepril, conivaptan, fenoldopam mesylate, or mirtazapine)
4. Subjects having taken an investigational drug within 30 days preceding randomization on Day 0
5. Subjects taking medications or having concomitant illnesses likely to confound endpoint assessments, including taking approved (ie, marketed) therapies for the purpose of affecting PKD cysts such as tolvaptan, somatostatin agonists (ie, octreotide, sandostatin), Rapamune (sirolimus), anti-sense RNA therapies, other vasopressin antagonists (eg, OPC-31260 [mozavaptan] and Vaprisol® [conivaptan]) or agonists (eg, desmopressin), and cyst reduction surgery
6. Subjects on antihypertensives that have not been on the same antihypertensive regimen for at least 30 days prior to the first dose of IMP
7. Subjects having contraindications to, or interference with, MRI assessments
8. Subjects with a history of serious mental disorders that, in the opinion of the investigator, would exclude the subject from participating in this trial
9. Subjects with previous exposure to tolvaptan

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, M.D., Ph.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (35):
- United States (35):
  - Otsuka Investigational Site, Huntsville, Alabama
  - Otsuka Investigational Site, Mobile, Alabama
  - Otsuka Investigational Site, Peoria, Arizona
  - Otsuka Investigational Site, Tempe, Arizona
  - Otsuka Investigational Site, Los Angeles, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site 2, Aurora, Colorado
  - Otsuka Investigational Site, Aurora, Colorado
  - Otsuka Investigational Site, Denver, Colorado
  - Otsuka Investigational Site, New Haven, Connecticut
  - Otsuka Investigational Site, Jacksonville, Florida
  - Otsuka Investigational Site, Melbourne, Florida
  - Otsuka Investigational Site, Atlanta, Georgia
  - Otsuka Investigational Site, Augusta, Georgia
  - Otsuka Investigational Site, Peoria, Illinois
  - Otsuka Investigational Site, Mishawaka, Indiana
  - Otsuka Investigational Site, Kansas City, Kansas
  - Otsuka Investigational Site, Paducah, Kentucky
  - Otsuka Investigational Site, Shreveport, Louisiana
  - Otsuka Investigational Site, Baltimore, Maryland
  - Otsuka Investigational Site, Rockville, Maryland
  - Otsuka Investigational Site, Boston, Massachusetts
  - Otsuka Investigational Site, Detroit, Michigan
  - Otsuka Investigational Site, Rochester, Minnesota
  - Otsuka Investigational Site, Voorhees Township, New Jersey
  - Otsuka Investigational Site, Buffalo, New York
  - Otsuka Investigational Site, Chapel Hill, North Carolina
  - Otsuka Investigational Site, Cleveland, Ohio
  - Otsuka Investigational Site, Bethlehem, Pennsylvania
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Anderson, South Carolina
  - Otsuka Investigational Site, Nashville, Tennessee
  - Otsuka Investigational Site, Arlington, Texas
  - Otsuka Investigational Site, Mission, Texas
  - Otsuka Investigational Site, Charlottesville, Virginia

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 177 participants at 41 trial states in the United States.
Pre-assignment Details: Participants entered a screening period within 4 weeks of being randomized (1:1:1:1) to one of four treatment groups. 178 is the number of subjects who enrolled due to informed consent, 177 is the number of subjects who were assigned to each treatment group.
Groups:
- Tolvaptan Modifed Release (MR) 50 mg: Tolvaptan MR 50 mg capsule and 2 placebo immediate release (IR) tablets (morning) and 1 placebo IR tablet (evening)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan MR 80 mg: Tolvaptan MR 80 mg capsule and 2 placebo immediate release (IR) tablets (morning) and 1 placebo IR tablet (evening)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan Immediate Release (IR) 60/30 mg: Two tolvaptan IR 30-mg tablets and 1 placebo MR capsule (morning) and 1 tolvaptan IR 30-mg tablet (evening)
  Tolvaptan IR: 60/30 mg capsules
  Placebo: tablet
- Placebo: Placebo MR capsule and 2 placebo IR tablets (morning) and 1 placebo IR tablet (evening)
  Placebo: tablet
Period: Overall Study
Arm/Group | Tolvaptan Modifed Release (MR) 50 mg | Tolvaptan MR 80 mg | Tolvaptan Immediate Release (IR) 60/30 mg | Placebo
Started | 45 | 45 | 44 | 43
Completed | 42 | 40 | 42 | 39
Not Completed | 3 | 5 | 2 | 4
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 2
Not completed — Participant met withdrawal criteria | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized to treatment.
Groups:
- Tolvaptan MR 50 mg: Tolvaptan MR 50 mg capsule and 2 placebo IR tablets (morning) and 1 placebo IR tablet (evening)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan MR 80 mg: Tolvaptan MR 80 mg capsule and 2 placebo IR tablets (morning) and 1 placebo IR tablet (evening)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan IR 60/30 mg: Two tolvaptan IR 30-mg tablets and 1 placebo MR capsule (morning) and 1 tolvaptan IR 30-mg tablet (PM)
  Tolvaptan IR: 60/30 mg capsules
  Placebo: tablet
- Placebo: Placebo MR capsule and 2 placebo IR tablets (evening) and 1 placebo IR tablet (morning)
  Placebo: tablet
- Total: Total of all reporting groups
Arm/Group | Tolvaptan MR 50 mg | Tolvaptan MR 80 mg | Tolvaptan IR 60/30 mg | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 44 | 43 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.1) | 35.8 (7.9) | 32.2 (7.6) | 33.9 (8.1) | 34.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 20 | 23 | 84
  Male | 27 | 22 | 24 | 20 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Kidney Volume (TKV) at Week 3
Description: The primary endpoint was percent change from baseline in TKV at Week 3. Total kidney volume is an important measure of disease progression. A 3-week time point is adequate to assess acute effects on kidney cyst shrinkage.
Time Frame: Baseline to Week 3
Population: Participants who were randomized and had baseline and post-baseline observations in the total renal volume.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Tolvaptan MR 50 mg: Tolvaptan MR 50 mg capsule and 2 placebo IR tablets (AM) and 1 placebo IR tablet (PM)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan MR 80 mg: Tolvaptan MR 80 mg capsule and 2 placebo IR tablets (AM) and 1 placebo IR tablet (PM)
  Tolvaptan MR: 50/80 mg capsules
  Placebo: tablet
- Tolvaptan IR 60/30 mg: Two tolvaptan IR 30-mg tablets and 1 placebo MR capsule (AM) and 1 tolvaptan IR 30-mg tablet (PM)
  Tolvaptan IR: 60/30 mg capsules
  Placebo: tablet
- Placebo: Placebo MR capsule and 2 placebo IR tablets (AM) and 1 placebo IR tablet (PM)
  Placebo: tablet
Arm/Group | Tolvaptan MR 50 mg | Tolvaptan MR 80 mg | Tolvaptan IR 60/30 mg | Placebo
Number analyzed (Participants) | 41 | 43 | 41 | 39
Percentage change | -2.46 (4.40) | -2.55 (3.85) | -1.17 (4.52) | 0.09 (5.31)
Statistical Analysis 1: Comparison: Tolvaptan MR 50 mg vs Tolvaptan MR 80 mg vs Tolvaptan IR 60/30 mg vs Placebo; Hierarchical tests were used to control the type I error in the primary analysis. They are given in the following order: 1. Pooled tolvaptan treatment groups (IR and MR) versus placebo; 2. Tolvaptan MR 80 mg versus placebo; 3. Tolvaptan MR 50 mg versus placebo; 4. Tolvaptan IR 60/30 mg versus placebo; Test type: Superiority or Other; p = 0.0127, ANCOVA; Ratio of geometric means = 0.98, 95% CI 2-sided [0.96 to 1.00]
Statistical Analysis 2: Comparison: Tolvaptan MR 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0108, ANCOVA; Ratio of geometric means = 0.97, 95% CI 2-sided [0.95 to 0.99]
Statistical Analysis 3: Comparison: Tolvaptan MR 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0155, ANCOVA; Ratio of geometric means = 0.98, 95% CI 2-sided [0.96 to 1.00]
Statistical Analysis 4: Comparison: Tolvaptan IR 60/30 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2417, ANCOVA; Ratio of geometric means = 0.99, 95% CI 2-sided [0.97 to 1.01]

2. Secondary Outcome: Change From Baseline in Total Score of the Autosomal Dominant Polycystic Kidney Disease Urinary Impact Scale (ADPKD-UIS)
Description: The ADPKD-UIS was a self-administered questionnaire designed to measure ADPKD-related urinary symptoms in participants with ADPKD. This instrument contained 11 items in 3 domains (Urinary Frequency, Urinary Urgency, and Nocturia). Each item was scored using a scale of 1 to 5 (a higher score indicated increased difficulty/extremely bothered). The maximum total score is 55; 1: not difficult/not bothered at all; 55: extremely difficult/extremely bothered.
Time Frame: Baseline to Week 8
Population: Participants who were randomized and had baseline and post-baseline observations in the total renal volume.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Tolvaptan MR 50 mg | Tolvaptan MR 80 mg | Tolvaptan IR 60/30 mg | Placebo
Number analyzed (Participants) | 39 | 40 | 42 | 38
Unit on a scale
  Urinary Frequency | 0.74 (0.94) | 0.82 (0.83) | 0.99 (0.78) | 0.10 (0.35)
  Urinary Urgency | 0.69 (0.96) | 0.66 (0.77) | 1.01 (0.95) | 0.05 (0.30)
  Nocturia | 0.97 (1.28) | 1.15 (0.89) | 1.36 (1.12) | 0.11 (0.59)
Statistical Analysis 1: Comparison: Tolvaptan MR 50 mg vs Placebo; Urinary Frequency; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.31 to 0.99]
Statistical Analysis 2: Comparison: Tolvaptan MR 80 mg vs Placebo; Urinary Frequency; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [0.40 to 1.08]
Statistical Analysis 3: Comparison: Tolvaptan IR 60/30 mg; Urinary Frequency; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [0.58 to 1.25]
Statistical Analysis 4: Comparison: Tolvaptan MR 50 mg vs Placebo; Urinary Urgency; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.30 to 1.01]
Statistical Analysis 5: Comparison: Tolvaptan MR 80 mg vs Placebo; Urinary Urgency; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.29 to 1.01]
Statistical Analysis 6: Comparison: Tolvaptan IR 60/30 mg vs Placebo; Urinary Urgency; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [0.63 to 1.34]
Statistical Analysis 7: Comparison: Tolvaptan MR 50 mg vs Placebo; Nocturia; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.42 to 1.30]
Statistical Analysis 8: Comparison: Tolvaptan MR 80 mg vs Placebo; Nocturia; Test type: Superiority or Other; p < 0.0001, ANCOVA; Median Difference (Final Values) = 1.07, 95% CI 2-sided [0.63 to 1.51]
Statistical Analysis 9: Comparison: Tolvaptan IR 60/30 mg vs Placebo; Nocturia; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [0.80 to 1.66]

3. Secondary Outcome: Percent Change From Baseline in TKV at Week 8.
Description: Total kidney volume is an important measure of disease progression. A 3-week time point is adequate to assess acute effects on kidney cyst shrinkage.
Time Frame: Baseline to Week 8
Population: The core patient population for all efficacy analyses was based on the intent-to-treat (ITT) population which consisted of all randomized participants who take at least one dose of study drug. Observed Cases (OC) dataset within treatment period was defined as the data observed at study specified visits while subjects are taking study drug.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Tolvaptan MR 50 mg | Tolvaptan MR 80 mg | Tolvaptan IR 60/30 mg | Placebo
Number analyzed (Participants) | 20 | 22 | 21 | 24
Percentage change | -2.04 (3.87) | -2.02 (3.54) | -0.08 (7.31) | 2.13 (7.99)
Statistical Analysis 1: Comparison: Tolvaptan MR 50 mg vs Tolvaptan MR 80 mg vs Tolvaptan IR 60/30 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0209, ANCOVA; Ratio of geometric means = 0.97, 95% CI 2-sided [0.94 to 0.99]
Statistical Analysis 2: Comparison: Tolvaptan MR 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0287, ANCOVA; Ratio of geometric means = 0.96, 95% CI 2-sided [0.93 to 1.00]
Statistical Analysis 3: Comparison: Tolvaptan MR 50 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0298, ANCOVA; Ratio of geometric means = 0.96, 95% CI 2-sided [0.93 to 1.00]
Statistical Analysis 4: Comparison: Tolvaptan IR 60/30 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2306, ANCOVA; Ratio of geometric means = 0.98, 95% CI 2-sided [0.94 to 1.01]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent, throughout the 8 week treatment period and for 7 days after the last dose of study medication.
Description: Safety analysis set consisted of all participants who took at least one dose of study medication. Serious adverse events, non-serious adverse events, and deaths were analyzed using safety analysis population.
Arm/Group | Tolvaptan MR 50 mg | Tolvaptan MR 80 mg | Tolvaptan IR 60/30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44 | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/45 | 1/44 | 1/44 | 1/42
Other Adverse Events (participants affected / at risk) | 27/45 | 25/44 | 32/44 | 18/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan MR 50 mg (N=45) | Tolvaptan MR 80 mg (N=44) | Tolvaptan IR 60/30 mg (N=44) | Placebo (N=42)
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan MR 50 mg (N=45) | Tolvaptan MR 80 mg (N=44) | Tolvaptan IR 60/30 mg (N=44) | Placebo (N=42)
Dry mouth (Gastrointestinal disorders) | 7 | 7 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 4
Fatigue (General disorders) | 3 | 2 | 6 | 1
Thirst (General disorders) | 15 | 15 | 19 | 6
Polydipsia (Metabolism and nutrition disorders) | 7 | 6 | 5 | 2
Headache (Nervous system disorders) | 1 | 1 | 7 | 1
Nocturia (Renal and urinary disorders) | 14 | 14 | 18 | 3
Pollakuria (Renal and urinary disorders) | 8 | 9 | 12 | 3
Polyuria (Renal and urinary disorders) | 11 | 11 | 13 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 1 | 2 | 3
Hypertension (Vascular disorders) | 2 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center may publish study results but ≥ 60 days prior to any public presentation, a copy is sent to Sponsor for review and Center can delay publication for 60 days to permit Sponsor to protect its intellectual property rights or confidential information contained within the publication. The first publication is a joint publication, if Center is part of a multi-center study. Center is free to publish, if there is no multi-center publication within 18 months of completion/ termination of study.